CLINICAL TRIAL: NCT05453266
Title: Arthroscopic Rotator Cuff Repair Performed With Intraarticular Tranexamic Acid. Could it Provide Improved Visual Clarity and Less Post-operative Pain? A Prospective, Double Blind, Randomized Study of 63 Patients
Brief Title: Arthroscopic Rotator Cuff Repair Performed With Intraarticular Tranexamic Acid Could it Provide Improved Visual Clarity and Less Post-operative Pain? A Prospective, Double Blind, Randomized Study of 64 Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florence Nightingale Hospital, Istanbul (Other)
Responsible Party: Principal Investigator, Celaleddin BILDIK, Principal Investigator, Florence Nightingale Hospital, Istanbul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13.02.2020/009
Record Dates: First submitted 2022-06-28; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Rupture; Tranexamic Acid; Shoulder Arthroscopy; Visual Clarity
Keywords: Rotator cuff tear; Rotator cuff rupture; Tranexamic acid; Shoulder arthroscopy; Visual clarity
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TXA Group (Active Comparator): Patients with rotator cuff tear, operated arthroscopically under intraarticularly applied tranexamic acid in arthroscopic irrigation solution.
  Interventions: Procedure: Application of Tranexamic acid in arthroscopic irrigation solution
- Control group (Placebo Comparator): Patients with rotator cuff tear, operated arthroscopically without intraarticularly applied tranexamic acid in arthroscopic irrigation solution.
  Interventions: Procedure: No application of Tranexamic acid in arthroscopic irrigation solution

INTERVENTIONS:
Procedure: Application of Tranexamic acid in arthroscopic irrigation solution — Application of Tranexamic acid in arthroscopic irrigation solution
  Arms: TXA Group
Procedure: No application of Tranexamic acid in arthroscopic irrigation solution — No application of Tranexamic acid in arthroscopic irrigation solution
  Arms: Control group

SUMMARY:
Shoulder arthroscopy is widely used for treatment of different shoulder pathologies. Visual clarity is essential for successful and safe surgery. The aim of present study is to determine whether intraarticular use of tranexamic acid (TXA) in surgery fluid can improve visual clarity and early postoperative pain.

DETAILED DESCRIPTION:
Patients and Methods After obtaining institutional review board approval (Istanbul Yeni Yuzyil University, Nr: 13.02.2020/009) together with the registry to ClinicalTrials.gov, patients were prospective enrolled in this observational study, which was designed as double-blind, placebo-controlled and randomized.

Inclusion criteria were defined as: being older than 18 years of age, having an MRI confirmed rotator cuff rupture with a history of failure of conservative treatment of at least 6 months, being willing to participate to the clinical trial.

Patient Selection Exclusion criteria were defined as: patients with a history of coagulopathy, deep venous thrombosis, tendency to thrombotic events, patients under anti-coagulant therapy, patients with inferior vena cava filter, patients with abnormal prothrombin time-activated partial thromboplastin time-bleeding time, patients with a history of cardiac/renal/hepatic disease, patients with a diagnosis of TXA allergy, patients with an acute RCT, having been treated conservatively for less than 6 months, being under the age of 18. Table 1.

As a result of the inclusion/exclusion criteria, 42 patients (14 had acute RCT, 12 were receiving anti-coagulant therapy, 9 had history of cardiac/hepatic/renal disease, 5 had abnormal PT-aPTT value at the time of the diagnosis, 2 had received conservative treatments for less than 6 months for RCR) were excluded from 105 patients, who were eligible and were willing to participate. The remaining 63 patients were enrolled in the study. Table 2 (Flowchart). All patients provided informed consents, so that their pre-operative, intra-operative and post-operative data including imaging studies and arthroscopic images could be used for publication by concealing their identity.

Randomization By using computer based randomization software acquired from random.org, patients were randomized into two groups comprising a TXA group (n=32, 24M, 8F) (TXA Group) and a control group (n=31, 22M,9F) (Control Group), while group information was neither shared with patients nor with the operating surgeon as a result of double-blind nature of the study.

Double-blinded preparation of the Irrigation Solutions To conduct a double-blinded, randomized control study, arthroscopic irrigation solutions (normal saline) of 3 liters were prepared by an operating nurse, while 250 mg TXA was injected into irrigation solutions of Group 1, and irrigation solutions of Group 2 were left TXA-free without any injection.

Surgical Procedures All procedures were performed under general anesthesia in beach-chair position by the same surgeon (C.B.) by following the exact same surgical steps in the exact same sequence irrespective of the patient's assignment to TXA group or control group. The surgical procedure comprised thorough evaluation of the glenohumeral joint, together with the rotator interval. In case of a degenerative biceps tendon, a biceps tenotomy was undertaken (TXA Group: 28 patients, Control Group: 26 patients). The repair of supraspinatus tendon was undertaken by utilizing single-row technique. A pressure-controlled pump was used to keep the pressure of the irrigation solution constantly at 50 mmHg. When visibility was decreased as a result of hemorrhage, the pressure was increased by 20 mmHg by using the flush option of the device. During the operation, mean arterial pressure was recorded by the anesthesiologist.

Assessment of Intra-Operative Arthroscopic Visual Clarity and Secondary Outcome Parameters Single surgeon (CB) rated arthroscopic visual score (AVS) similar to the grading system used by van Montfoort21 was used to evaluate intra-operative clarity. AVS was composed of five grades: Grade I: I had no disruption of visual clarity due to bleeding.

Grade II: I had mild disruption of visual clarity due to bleeding. Grade III: I had moderate disruption of visual clarity due to bleeding. Grade IV: I had severe disruption of visual clarity due to bleeding. Grade V: As a result of extreme disruption of visual clarity due to bleeding, I had to convert to open surgery.

AVS score for every patient was calculated as the following: The video of the operation was watched by the operating surgeon (CB) after the surgery and at every 15 minutes, a score of AVS was recorded. At the end, the average score for every single patient was calculated.

Pain was evaluated by using visual analogue scale (VAS) post-operative 8th, 24th and 48th hour.

Patients' mean arterial pressures (MAP) and total duration of operations were recorded.

All of the average aforementioned data of the two groups were compared. Post-operative Patient Management Patients were applied abduction brace after the operation and they were advised to limit the active shoulder range of motion together with abduction during their stay in the hospital.

Pain management was performed by 500 mg paracetamol injection at every 8 hours and intramuscular injection of ketorolac at 24 hours. Patients were discharged at the second post-operative day, when they were confirmed to be stable with tolerable pain.

Statistical method To calculate the sample size, G-Power software (gpower.hhu.de, v 3.1.9.4) was used, while a statistical power (1-ß), alpha error and impact value were calculated as 0.8, 0.05 and 0.8 respectively. As a result of this priori power analysis model, at least 30 speciments were calculated to be required in each group, which was consistent with out design.

For the statistical analysis SPSS software (Version 25.0; SPSS Inc, Chicago, IL, USA) was used. Data are expressed as mean +/- SD (standard deviation). The cohort and the variables were tested for normal distribution and data normality was confirmed by Shapiro-Wilk test. Age, sex, surgery time, mean arterial blood pressure, surgical visaualization score, AVS and postoperative pain scores were compared between groups. Demographic characteristics of the patients were analyzed using descriptive statistics analysis methods, with mean and standard deviation. Normality analysis was made with different methods including histogram, kurtosis and skewness test. Independent sample t-test was used to compare the difference between groups. Analysis of postoperative pain scores at different time points scores within the groups at different time points was made with repeated measures ANOVA test. Results were reported at a 95% confidence interval, and P values <0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* being older than 18 years of age,
* having an MRI confirmed rotator cuff rupture with a history of failure of conservative treatment of at least 6 months,
* being willing to participate to the clinical trial.

Exclusion Criteria:

* patients with a history of coagulopathy, deep venous thrombosis, tendency to thrombotic events,
* patients under anti-coagulant therapy,
* patients with inferior vena cava filter,
* patients with abnormal prothrombin time-activated partial thromboplastin time-bleeding time,
* patients with a history of cardiac/renal/hepatic disease,
* patients with a diagnosis of TXA allergy,
* patients with an acute RCT, having been treated conservatively for less than 6 months,
* being under the age of 18

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Arthroscopic Visual Clarity | Intra-operatively
  Effect of TXA in arthroscopic irrigation solution to Arthroscopic Visual Clarity

SECONDARY OUTCOMES:
Post-operative Pain Evaluation | Up to the 2nd post-operative day
  Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Ataşehir Florence Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the IPD.